CLINICAL TRIAL: NCT00558792
Title: A Phase II Multicenter Randomized Double Blind Dose Finding Study of Iopamidol Injection 370 in Multidetector Computed Tomographic Angiography (MDCTA) in Patients With Suspected Coronary Artery Stenosis
Brief Title: Coronary MDCTA With Iopamidol Injection 370
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP 108; NCT00558792 (Registry Identifier: clinicaltrials.gov)
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isovue 370, 70 mL (Experimental): iopamidol injection 370, 70 mL
  Interventions: Drug: Isovue 370, 70 mL
- Isovue 370, 80 mL (Experimental): iopamidol injection 370, 80 mL
  Interventions: Drug: Isovue 370, 80 mL
- Isovue 370, 90 mL (Experimental): iopamidol injection 370, 90 mL
  Interventions: Drug: Isovue 370, 90 mL

INTERVENTIONS:
Drug: Isovue 370, 70 mL — 70 mL of iopamidol injection 370 injected at a rate of >=4 mL/second
  Other Names: Isovue
  Arms: Isovue 370, 70 mL
Drug: Isovue 370, 80 mL — 80 mL of iopamidol injection 370 injected at a rate of >=4 mL/second
  Other Names: Isovue
  Arms: Isovue 370, 80 mL
Drug: Isovue 370, 90 mL — 90 mL of iopamidol injection 370 injected at a rate of >=4 mL/second
  Other Names: Isovue
  Arms: Isovue 370, 90 mL

SUMMARY:
Determine the validity and compare the visualization of arterial segments obtained with 3 doses of iopamidol to determine dose for further investigation in future trials.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* At least 30 years of age
* Weight less than 250 lbs
* Known or suspected coronary artery disease and suspected to have significant coronary artery stenosis
* Undergo MDCTA scan
* Undergo coronary angiography within 2 weeks of MDCTA scan

Exclusion Criteria:

* Hx of hypersensitivity to iodinated contrast agents
* Known or suspected hyperthyroidism or pheochromocytoma
* Renal impairment
* History of coronary artery stent placement or bypass grafts
* Unstable
* Pregnant or lactating

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiefen Yao, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from December 2007 to December 2009 in 17 investigational sites across the United States of America (USA), 2 investigational sites in Canada and 2 investigational sites in Italy. A blinded read of the images obtained during the study was performed in May 2010.
Pre-assignment Details: This was a Phase II, multicenter, prospective, double-blind, randomized, parallel-group comparison of 3 doses of iopamidol injection 370 when used for coronary MDCTA.
Period: Overall Study
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Started | 68 | 63 | 60
Completed | 68 | 63 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL | Total
Number analyzed (Participants) | 68 | 63 | 60 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 49 | 42 | 144
  >=65 years | 15 | 14 | 18 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.85) | 57.7 (8.54) | 58.7 (9.25) | 58.0 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 21 | 73
  Male | 43 | 36 | 39 | 118
Region of Enrollment [Number; unit: participants]
  United States | 55 | 50 | 48 | 153
  Canada | 11 | 10 | 10 | 31
  Italy | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Quality of Visualization of Coronary Arteries, Off-Site Reader 1
Description: For all technically adequate coronary artery segments, each reader was to assess whether each segment was visualized to a quality that was adequate for accurate diagnosis of the presence and severity of stenosis. An adequate quality for the accurate diagnosis of the presence and severity of coronary artery stenosis was comprised of 2 basic features: 1) no more than mild blurring of the spatial distinction between the vessel wall and lumen, and 2) a readily visible distinction in image contrast between calcified plaque, enhanced vessel lumen, and uncalcified vessel wall or plaque.
Time Frame: Immediately post dose
Measure: Number; unit: Segments Visualized Accurately
Units Other Than Participants: Segments Present & Technically Adequate
Groups:
- Isovue 370, 70 mL: Patients received a randomized total dose of Iopamidol injection 370, which could be 70, 80, or 90 milliliters (mL), at a rate of >4 mL per second (/sec), followed by a 40 mL saline flush, administered at the same injection rate.
- Isovue 370, 80 mL; Isovue 370, 90 mL: Patients received a randomized total dose of Iopamidol injection 370, which could be 70, 80, or 90 mL, at a rate of >4 mL/sec, followed by a 40 mL saline flush, administered at the same injection rate.
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 68 | 62 | 60
Number analyzed (Segments Present & Technically Adequate) | 963 | 865 | 848
Segments Visualized Accurately | 949 | 842 | 841
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.0099, Chi-squared

2. Primary Outcome: Diagnostic Quality of Visualization of Coronary Arteries, Off-Site Reader 2
Description: as for outcome 1
Time Frame: Immediately post dose
Measure: Number; unit: Segments Visualized Accurately
Units Other Than Participants: Segments
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 68 | 62 | 60
Number analyzed (Segments) | 1042 | 950 | 927
Segments Visualized Accurately | 1032 | 924 | 927
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Primary Outcome: Diagnostic Quality of Visualization of Coronary Arteries, Off-Site Reader 3
Description: as for outcome 1
Time Frame: Immediately post dose
Measure: Number; unit: Segments Visualized Accurately
Units Other Than Participants: Segments Present & Technically Adequate
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 68 | 62 | 60
Number analyzed (Segments Present & Technically Adequate) | 925 | 826 | 817
Segments Visualized Accurately | 925 | 824 | 817
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.1212, Chi-squared

4. Secondary Outcome: Number of Participants Who Experienced Adverse Events With Incidence of 5% or Greater
Description: Participants who received investigational product (iopamidol injection) and experienced an adverse event (AE). See Adverse Events module for further details.
Time Frame: up to 72 hours post dose
Measure: Number; unit: Participants who Experienced AE(s)
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 68 | 63 | 60
Participants who Experienced AE(s) | 15 | 14 | 13

5. Primary Outcome: Contrast Density (CD) Measurements, Off-Site Reader 1
Description: For this assessment, each off-site reader was to place regions of interest (ROIs) into the lumens of the mid-portion of the left main coronary artery (LM) (segment number 5), and into the mid-portion of segment number 1 of the right coronary artery (RCA). The mean Hounsfield Units levels and standard deviations (SD) for those 2 ROIs were to be recorded by the reader.
Time Frame: Immediately post dose
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 67 | 58 | 59
Hounsfield Units | 372.806 (90.5842) | 398.255 (82.3593) | 418.197 (97.4072)
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.0200, ANOVA

6. Primary Outcome: Contrast Density (CD) Measurements, Off-Site Reader 2
Description: as for outcome 5
Time Frame: Immediately post dose
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 67 | 58 | 58
Hounsfield Units | 364.784 (78.2154) | 396.291 (85.7038) | 413.665 (86.0972)
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.0044, ANOVA

7. Primary Outcome: Contrast Density (CD) Measurements, Off-Site Reader 3
Description: as for outcome 5
Time Frame: Immediately post dose
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 64 | 58 | 57
Hounsfield Units | 363.071 (85.7795) | 383.841 (96.8142) | 406.206 (91.9117)
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.0371, ANOVA

8. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 1 - Sensitivity
Description: For each technically adequate coronary artery, the readers assessed or excluded the presence of coronary artery stenoses. If more than one stenosis was present in a single vessel, the readers recorded the most significant stenosis. Based on a match or mismatch between computed tomographic angiography (CTA) and coronary angiography as assessed by the adjudicator, each vessel diagnosis by CTA was defined as true negative (TN), false positive (FP), false negative (FN), or true positive (TP) based on coronary angiography findings. Technical inadequacy by multi-detector CTA was counted as FN or FP depending on the diagnostic results from conventional angiography. The percentage (%) of sensitivity [TP/(TP+FN)] is presented.
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Sensitivity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Sensitivity (%) | 63.6 | 65.5 | 77.8
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.2758, Chi-squared — Study was not powered for diagnostic performance analyses. Sample size was based on quality of visualization of coronary artery segments; Difference in Sensitivity between Doses = 14.1, 95% CI 2-sided [-11.4 to 39.6]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.3102, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 12.3, 95% CI 2-sided [-11.1 to 35.6]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.8893, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 1.9, 95% CI 2-sided [-24.6 to 28.4]

9. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 1 - Specificity
Description: For each technically adequate coronary artery, the readers assessed or excluded the presence of coronary artery stenoses. If more than one stenosis was present in a single vessel, the readers recorded the most significant stenosis. Based on a match or mismatch between computed tomographic angiography (CTA) and coronary angiography as assessed by the adjudicator, each vessel diagnosis by CTA was defined as true negative (TN), false positive (FP), false negative (FN), or true positive (TP) based on coronary angiography findings. Technical inadequacy by multi-detector CTA was counted as FN or FP depending on the diagnostic results from conventional angiography. The percentage (%) of specificity [TN/(TN+FP)] is presented.
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Specificity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Specificity (%) | 98.3 | 95.2 | 96.6
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.2511, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -1.7, 95% CI 2-sided [-4.7 to 1.3]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.4985, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = 1.3, 95% CI 2-sided [-2.6 to 5.3]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.0693, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -3.1, 95% CI 2-sided [-6.5 to 0.4]

10. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 2 - Sensitivity
Description: as for outcome 8
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Sensitivity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Sensitivity (%) | 68.2 | 79.3 | 66.7
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.9104, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = -1.5, 95% CI 2-sided [-27.9 to 24.8]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.2857, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = -12.6, 95% CI 2-sided [-35.7 to 10.5]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.3664, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 11.1, 95% CI 2-sided [-13.3 to 35.5]

11. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 2 - Specificity
Description: as for outcome 9
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Specificity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Specificity (%) | 94.5 | 92.1 | 90.7
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.1322, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specifcity between Doses = -3.7, 95% CI 2-sided [-8.7 to 1.2]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.6381, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -1.3, 95% CI 2-sided [-6.9 to 4.2]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.3217, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -2.4, 95% CI 2-sided [-7.2 to 2.4]

12. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 3 - Sensitivity
Description: as for outcome 8
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Sensitivity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Sensitivity (%) | 59.1 | 62.1 | 66.7
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.5843, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 7.6, 95% CI 2-sided [-19.6 to 34.7]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.7197, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 4.6, 95% CI 2-sided [-20.5 to 29.7]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.8292, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Sensitivity between Doses = 3.0, 95% CI 2-sided [-24.1 to 30.1]

13. Primary Outcome: Validity (Sensitivity and Specificity), Off-Site Reader 3 - Specificity
Description: as for outcome 9
Time Frame: Immediately post dose
Population: Number of participants with significant disease (>50% stenosis)
Measure: Number; unit: Specificity (%)
Units Other Than Participants: Vessels
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Number analyzed (Participants) | 65 | 55 | 58
Number analyzed (Vessels) | 257 | 218 | 232
Specificity (%) | 94.9 | 91.5 | 90.7
Statistical Analysis 1: Comparison: Isovue 370, 70 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.0888, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -4.2, 95% CI 2-sided [-9.0 to 0.7]
Statistical Analysis 2: Comparison: Isovue 370, 80 mL vs Isovue 370, 90 mL; Test type: Superiority or Other; p = 0.7796, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -0.8, 95% CI 2-sided [-6.4 to 4.8]
Statistical Analysis 3: Comparison: Isovue 370, 70 mL vs Isovue 370, 80 mL; Test type: Superiority or Other; p = 0.1662, Chi-squared — [p-value comment as in outcome 8, analysis 1]; Difference in Specificity between Doses = -3.4, 95% CI 2-sided [-8.2 to 1.5]

ADVERSE EVENTS:
Time Frame: Patients were monitored for any untoward medical occurrence from the time they signed the informed consent until 72 hours after the administration of iopamidol injection 370.
Description: Only those adverse events that were reported after the injection of iopamidol injection 370 are presented.
Arm/Group | Isovue 370, 70 mL | Isovue 370, 80 mL | Isovue 370, 90 mL
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/63 | 0/60
Other Adverse Events (participants affected / at risk) | 15/68 | 14/63 | 13/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isovue 370, 70 mL (N=68) | Isovue 370, 80 mL (N=63) | Isovue 370, 90 mL (N=60)
Feeling Hot (General disorders) | 6 (6) | 5 (5) | 5 (5)
Flushing (Vascular disorders) | 4 (4) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 7 (7) | 6 (6) | 2 (2)
Injection Site Erythema (General disorders) | 0 (0) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be presented during scientific symposia or published in a scientific journal only after review by Bracco in accordance with the guidelines set forth in the applicable publication or financial agreement.